CLINICAL TRIAL: NCT03778827
Title: A Center Based Randomized Controlled Trial of Pivotal Response Treatment for Preschoolers With Autism
Brief Title: A Center Based Study of Pivotal Response Treatment for Preschoolers With Autism
Acronym: PRT-C
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: John & Marcia Goldman Foundation (Unknown)
Responsible Party: Principal Investigator, Antonio Hardan, Professor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-49033
Record Dates: First submitted 2018-12-15; First posted 2018-12-19 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Autism Spectrum Disorder; Autism
Keywords: Pivotal Response Treatment
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Center-Based Pivotal Response Treatment (PRT-C) (Experimental): Intensive Center-Based Pivotal Response Treatment (PRT-C) will consist of a combination of one weekly 60-minute individual parent training session and 12 weekly hours ( 3 hours per day for 4 days per week) with the child in center-based therapy environment for a total of 13 weekly treatment hours.
  Interventions: Behavioral: Intensive Center-Based Pivotal Response Treatment (PRT-C)
- Delayed Treatment Group (DTG) (No Intervention): Delayed Treatment Group will consist of treatment as usual. At the end of controlled phase, participants in the DTG will be offered PRT-C in a preschool setting in an open-label fashion with a design similar to the double-blind phase.

INTERVENTIONS:
Behavioral: Intensive Center-Based Pivotal Response Treatment (PRT-C) — Intensive Center-Based Pivotal Response Treatment (PRT-C) will consist of a combination of weekly individual parent training sessions and center-based therapy for a total of 13 weekly treatment hours.
  Arms: Intensive Center-Based Pivotal Response Treatment (PRT-C)

SUMMARY:
The purpose of this study is to examine the effectiveness of pivotal response training (PRT) in an intensive center-based environment to treat social communication deficits in children with autism spectrum disorder (ASD).

DETAILED DESCRIPTION:
The purpose of this study is to examine the effectiveness of pivotal response training (PRT) in an intensive center-based preschool environment to treat social communication deficits in children with autism spectrum disorder (ASD). The study will compare Pivotal Response Treatment (PRT) to a delayed treatment group (DTG). PRT is a naturalistic behavioral intervention based on the principles of applied behavior analysis which has shown to be effective in treating the core deficits in children with ASD. The study will compare the combination of parent training with intensive center-based PRT (PRT-C) to a DTG and will include 44 children ages 2 to 3.11 years with ASD and social communication deficits.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autism Spectrum Disorder (ASD) based on clinical interview and Diagnostic and Statistical Manual, 5th edition (DSM-5) and confirmed using the Autism Diagnostic Interview Revised (ADI-R) and Autism Diagnostic Observation Schedule, 2nd edition (ADOS-2) or Childhood Autism Rating Scale (CARS-2); Diagnostic and Statistical Manual, 5th edition (DSM-5), and expert clinical opinion
* Boys and girls between 2 years and 3 years and 11 months
* Ability to participate in the testing procedures to the extent that valid standard scores can be obtained
* Stable treatment (e.g., applied behavior analysis (ABA), speech therapy, psychotropic medication(s) or biomedical intervention(s) for at least 1 month prior to baseline measurements with no anticipated changes during study participation
* Developmentally delayed with Mullen Scales of Early Learning (MSEL) or Developmental Profile (DP-4) composite score below 85 (1 Standard Deviation below the mean)
* Availability of at least one English-speaking parent who can consistently participate in parent training and research measures.

Exclusion Criteria:

* Current or lifetime diagnosis of severe psychiatric disorder (e.g., bipolar disorder, etc.)
* Presence of active medical problem (e.g., unstable seizure disorder or heart disease)
* Child primary language other than English
* Previous adequate trial of Pivotal Response Treatment
* More than 15 hours per week of in-home applied behavior analysis (ABA).

Ages: 2 Years to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Mean Change from baseline on the Social Responsiveness Scale-2 Total Score at 12 Weeks | Baseline and Week 12
Mean change from baseline on the Brief Observation of Communication Change (BOSCC) total score at 12 Weeks | Baseline and Week 12
Mean change from baseline on the frequency if the child's functional utterances on the structured lab observation at 12 Weeks | Baseline and Week 12

SECONDARY OUTCOMES:
Mean change from baseline on the Vineland Adaptive Behavior Scales 3rd Edition Socialization subscale at 12 Weeks | Baseline and Week 12
Mean change from baseline on the MacArthur-Bates Communication Development Inventory at 12 Weeks | Baseline and Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Y. Hardan, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No